CLINICAL TRIAL: NCT04210323
Title: Use of Shotblocker® in Subcutaneous Injecting in Chronic Spontaneous Urticaria Patients: Randomized Placebo Controlled Study
Brief Title: Shotblocker® Use in Subcutaneous Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Merve Kolcu, Assistant Professor, Director, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: omalizumab; subcutaneous; injection; ShotBlocker
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shotblocker group (Experimental): ShotBlocker® was used by an experienced registered nurse under the researcher supervision. The injection area gripped with ShotBlocker®, released after the drug administration and then the ShotBlocker® was removed. After injection, light pressure was applied to the injection area with dry cotton.
  Interventions: Device: ShotBlocker®
- Placebo group (Placebo Comparator): The smooth surface (opposite side) of the ShotBlocker® was placed in the injection area just before administration by an experience registered nurse and the drug was injected by holding it on the skin surface during the injection. The process was managed by the researcher.
  Interventions: Device: Placebo group
- Control group (No Intervention): Subcutaneous injection was performed with normal subcutaneous drug administration steps by an experienced registered nurse and no additional method was applied. The application process of each patient was managed by the researcher.

INTERVENTIONS:
Device: ShotBlocker® — The injection area gripped with ShotBlocker®, released after the drug administration and then the ShotBlocker® was removed. After injection, light pressure was applied to the injection area with dry cotton.
  Arms: Shotblocker group
Device: Placebo group — The smooth surface (opposite side) of the ShotBlocker® was placed in the injection area just before administration by an experience registered nurse and the drug was injected by holding it on the skin surface during the injection. The process was managed by the researcher.
  Other Names: The smooth surface of the ShotBlocker®
  Arms: Placebo group

SUMMARY:
Aim: The aim of this study was to investigate the effect of subcutaneous injection with ShotBlocker® on patients with chronic spontaneous urticaria.

Background: In chronic diseases such as CSU, after subcutaneous injection, problems such as pain, ecchymosis and hematoma may arise due to the injection technique. This may lead to tissue loss at the injection site subsequent injections of subcutaneously administered omalizumab every twenty-eight days and increase the stress level.

Design: Randomized placebo controlled. Methods: Data were collected between June-November 2018 by including 90 patients out of 125 patients with Chronic Spontaneous Urticaria in Dermatology Clinic, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey. Patients were divided into three groups as intervention, control and shotblocker group. Patients in the placebo group were administered with the reverse side of ShotBlocker® during subcutaneous injection, and no intervention was performed in the control group. The group using ShotBlocker® for subcutaneous injection was compared with the placebo and control groups.

DETAILED DESCRIPTION:
In chronic diseases such as CSU, after subcutaneous injection, problems such as pain, ecchymosis and hematoma may arise due to the injection technique. This may lead to tissue loss at the injection site subsequent injections of subcutaneously administered omalizumab every twenty-eight days and increase the stress level . It is stated in the literature that complications may be reduced significantly with appropriate technique in subcutaneous injection applications.

For this purpose, "ShotBlocker® (Bionix, Toledo, Ohio) was developed for subcutaneous and intramuscular injection applications. ShotBlocker® is a drug-free, non-invasive plastic device that can be applied for all age groups. It simulates the smaller nerves at the injection site and briefly blocks the pain gate in the central nervous system and slows down A-delta signals. ShotBlocker® is quick and easy to use, does not require any preliminary preparation, and has not been previously reported side effects. A surface of the device has a plurality of blunt spots these directly in contact with the skin. It is reported that the injection pain is reduced by applying light pressure to the contacting area with a short, non-sharp 2 mm thick blunt tip. There is a gap in the middle of the device to display the injection site and injection is applied through this gap.

In most international studies, it has been found that subcutaneous and intramuscular injection with ShotBlocker® has a substantial impact on reducing pain levels. It has been found the limited number of studies have been published in Turkey in order to evaluate the effectiveness of ShotBlocker® devices in pain. In the literature review, there was not found any published research about the use of Shot Blocker® in patients with CSU who received regular subcutaneous injections.

With the results of this research, it is believed that an effective method can be presented to reduce the pain and anxiety related with subcutaneous injection and increase the level of satisfaction in CSU patients, and to contribute the development of patient care with safe practices.

ELIGIBILITY:
Inclusion Criteria:

* Communicative
* 18 years and older
* Body Mass Index (BMI) between 18.5-29.9 kg / m²
* CSU diagnosed
* Having regular subcutaneous omalizumab treatment
* Having not infection, scar tissue or incision on the posterior side of both upper arms and another parenteral treatment was not applied that side.
* Having not any haematological disease
* Volunteer to participate in the research

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Visual comparison scales | 60 minutes
  Visual Analog Scales (VAS) were used in order to determine the pain and satisfaction of the administration. The scale comprise of a 10 cm long horizontal line with descriptive expressions at both ends (0 cm: no pain / no satisfaction and 10 cm on the right end: unbearable pain / very satisfied). Participants were asked to mark the pain level on this line.

SECONDARY OUTCOMES:
The state-trait anxiety inventory form TX-I | 1 week
  STAI was developed by Spielberger et al. In 1970 to measure state (TX-I) and trait anxiety levels (TX-II), and was adapted to Turkish society in 1985 by Öner and Le Compte. The State-Trait Anxiety Scale (TX-I) used in this study is a Likert-type scale consisting of 20 questions to determine how an individual feel at a given time and under certain circumstances. Each question has four options; 10 items are the reverse items (1,2,5,8,10,11,15,16,19 and 20), the lowest score is 20 and the highest score is 80. A higher score indicates a high level of anxiety and a lower score indicates a low level of anxiety.
Visual comparison scales | 1 week
  Visual Analog Scales (VAS) were used in order to determine the pain and satisfaction of the administration. The scale comprise of a 10 cm long horizontal line with descriptive expressions at both ends (0 cm: no pain / no satisfaction and 10 cm on the right end: unbearable pain / very satisfied). Participants were asked to mark satisfaction level on this line.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No